CLINICAL TRIAL: NCT02745652
Title: Pulsed Magnetic Field Versus Ultrasound in Treatment of Postnatal Carpal Tunnel Syndrome: Randomized Control Trial on Female Egyptian Population
Brief Title: Carpel Tunnel Syndrome and Physical Therapy Modalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dr. Dalia Mohamed Kame, Associate Professor of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/001211
Record Dates: First submitted 2016-04-14; First posted 2016-04-20 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Carpal Tunnel Syndrome
Keywords: median nerve; wrist joint; carpal tunnel
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy | interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pulsed electromagnetic field (PEMF) (Experimental): patients in this group received the pulse electromagnetic field with frequency 50 Hz and intensity 80 gauss for 30 min.The patient was in sitting position, while the forearm was rested on the bed inside the solenoid in supination position
  Interventions: Device: pulsed electromagnetic field
- Therapeutic ultrasound (US) (Experimental): Pulsed mode US was applied over the volar surface of the forearm (the carpal tunnel area) 15 min per session with a frequency of 1 MHz and intensity of 1.0 W/cm2
  Interventions: Device: Therapeutic ultrasound

INTERVENTIONS:
Device: pulsed electromagnetic field — it is a magnetic device for magneto-therapy, it has an appliance, motorized bed, and applicable large solenoids which can be moved in 4 different positions according to the treatment area, and the additional small solenoid for hand treatment with 30 cm diameter
  Other Names: (PEMF)
  Arms: pulsed electromagnetic field (PEMF)
Device: Therapeutic ultrasound — Ultrasound is applied using a transducer or applicator that is in direct contact with the patient's skin. Gel is a medium which is used on all surfaces of the head to reduce friction and assist transmission of the ultrasonic waves
  Other Names: US
  Arms: Therapeutic ultrasound (US)

SUMMARY:
Carpel tunnel syndrome (CTS) is very common complain during pregnancy with high percentage to continue postnatal. Conservative treatment is more recommended in these cases. There are many physical therapy modalities proposed to treat CTS without knowing which modality is better than the other. So the aim of this study to compare the effect of two modalities in treating CTS in postnatal females.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is one of the most common peripheral nerve entrapment disorders in the upper limb. CTS is common during pregnancy especially in the third trimester as well, a significant percentage of females postnatal may still have some complaints up to at least 3 years postnatal.

Purpose: To compare the effect of pulsed magnetic field (PEMF) versus ultrasound (US) in treating patients with CTS. Forty postnatal female patients with idiopathic CTS were assigned randomly into two equal groups. One group received PEMF with nerve and tendon gliding exercises for the wrist 3 times for week for 4 weeks. The other group received US plus the same exercises. Pain level, sensory and motor distal latencies of the median nerve (MSDL and MMDL), sensory and motor conduction velocities of the median nerve (MSCV and MMCV), functional status scale and hand grip strength were assessed pre and post treatment

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate CTS
* Positive electro diagnostic findings: prolonged median motor distal latency (MMDL) above 4 ms, and below 6ms.
* Prolonged median sensory distal latency above 3.5 ms .
* Positive Phalen and Tinel test.
* Subjects scored pain intensity more than 5 in visual analogue scale (VAS).

Exclusion Criteria:

* severe cases with delayed motor distal latency > 6ms.
* Orthopedic or neurological disorders of neck or the upper limb as cervical radiculopathy.
* Pronator teres syndrome or double crush syndrome.
* Pre- existing CTS before their last pregnancy, current pregnancy.
* Diabetic neuropathy and Thoracic outlet syndrome.
* Wasting of thenar muscles, ulnar neuropathy.
* Rheumatoid arthritis, previous fractured carpal bone and previous surgery in the forearm especially transverse ligament release

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks change from the baseline scores
  it measured by the Visual Analogue Scale (VAS).It is considered a valid way of assessing pain

SECONDARY OUTCOMES:
Functional status scale | 4 weeks change from the baseline scores
  It is a part of the Carpal Tunnel Syndrome Questionnaire (CTSQ). it asks about eight functional activities as writing, buttoning of clothes, gripping of a telephone handle

IPD SHARING:
Plan to Share IPD: Yes
publication in a refereed journal